CLINICAL TRIAL: NCT02842905
Title: Examining the Impact of Physician Influence on Hearing Aid User Satisfaction and Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: NexGen Hearing Inc. (Unknown)
Responsible Party: Principal Investigator, Desmond A Nunez, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H15-01282
Record Dates: First submitted 2016-07-13; First posted 2016-07-25 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

ARMS (2):
- Control Group (Active Comparator): Fitting Audiologist completion of the Client Outcome Scale of Improvement at a post fitting follow up visit.
  Interventions: Other: Fitting Audiologist completion
- Test Group (Experimental): Participant's physician completion of the Client Outcome Scale of Improvement at a post fitting follow up visit.
  Interventions: Other: Participant's Physician completion

INTERVENTIONS:
Other: Fitting Audiologist completion — Phase II of the COSI (Client Oriented Scale of Improvement) questionnaire completed in a scheduled visit with the fitting Audiologist
  Arms: Control Group
Other: Participant's Physician completion — Phase II of the COSI (Client Oriented Scale of Improvement) questionnaire completed in a scheduled visit with the Participant's Physician
  Arms: Test Group

SUMMARY:
Most of us will experience some degree of hearing loss as we get older. It can affect one or both ears and without treatment causes difficulty with following conversations in the home or workplace. Audiologists are trained to diagnose and treat hearing loss and tinnitus problems. They also dispense, and fit hearing aids. Physicians do not provide or fit hearing aids directly, however they diagnose hearing loss and can recommend hearing aids amongst other treatments for hearing loss. It is undecided whether consulting with a physician in addition to an audiologist will improve user's satisfaction with hearing aids, compared to consulting with an audiologist alone.

The purpose of this study is to determine whether physician involvement (in addition to an audiologist) in the hearing aid fitting process improves users' satisfaction with hearing aids. The study utilizes questionnaires to assess satisfaction with hearing aids. Furthermore, participants decision to keep the purchased hearing aids will be recorded.

The study will take place in the clinics of family doctors, Otolaryngology (Ear) surgeons and audiologists. A hearing aid suitable for the needs of the participant will be fitted by an audiologist. In the first 21days after the fitting, participants will attend follow-up visits with the audiologists for adjustments to the hearing aids to best meet their specific listening needs. After 21 days, eligible participants will be allocated to either the Control or Test groups. Participants in both groups will be asked to describe the change in their hearing performance related to the use of hearing aids to their audiologist(Control) or Physician (Test) at a follow-up visit. At the study's final visit, participants will be asked to complete a satisfaction-based questionnaire.

The time taken to fit a hearing aid varies depending on the individual needs of the patient. It is estimated that at most 10 visits will be required over 90 days to complete the hearing aid fitting and study processes. These visits will be of 30 minutes duration on average, except for the initial and final visits which lasts for 45 minutes. A patient will spend a maximum of 330 minutes to complete the hearing aid fitting process, but only 25 minutes of this time will be specifically related to the study.

The study is intended to determine the satisfaction with hearing aids and consultations with health professionals.

DETAILED DESCRIPTION:
Description of study design This study seeks to determine if additional patient benefit is derived from involving the referring physician in the hearing aid fitting process using the Client Oriented Scale of Improvement (COSI) process. The COSI process is a well-known methodology that consists of two consecutive phases: Phase I is completed by the client with the Audiologist either at the time of initial hearing aid fitting or within 21 days thereafter. The patient is asked to list any specific listening environment/situations in which he/she would like to improve his/her hearing with the assistance of wearing hearing aids; Phase II occurs within days 22 to 76 from the day the hearing aid device is fitted and is also normally completed by the patient and the Audiologist. In this phase, the patient indicates any degree of change in the specific listening environment/situations he/she had previously listed (wearing the hearing aid).

Two methods will be used for study purposes to assess patient satisfaction with hearing aid use 77 to 90 days post fitting: (1) the validated SADL questionnaire described previously will be completed by the patient and (2) the number of hearing aids returned up to 90 days post initial fitting will be recorded.

The study will consist of two groups: a control group and a test group. Both groups will undergo Phase I of the COSI process with the fitting Audiologist. Patients in the control group will undergo Phase II of the COSI process as part of their follow up with the audiologist, whereas those in the test group will complete Phase II of the COSI process in a scheduled visit with their referring physician before further follow-up with the audiologist. Participants will be recruited from the investigating audiologists' clinics in Vancouver. The study involvement time for each participant will extend over a period of 90 days.

Routine Clinical Practice A complete hearing aid fitting takes place over the course of several clinic visits each on average 30-45 minutes in duration. These include the initial hearing test and consultation, actual fitting, and any subsequent post-fitting adjustments. During hearing evaluation and post-fitting follow-up sessions, a COSI questionnaire is used by audiologists as part of routine clinical practice to guide optimal hearing aid adjustment to meet the patient's listening needs.

Time schedule The time taken to fit a hearing aid varies depending on the needs of the patient. Very often clients over the age of 55 have problems with dexterity, memory and other health impairments that extend the length of individual consultations. Some patients require more clinic consultations than others. Anecdotally it is estimated that the maximal number of visits required to complete the hearing aid fitting process is 10 visits over 90 days. These visits on average will be of 30 minutes in duration except for the initial and final visits which lasts for 45 minutes. A patient will spend a maximum of 330 minutes to complete the hearing aid fitting process of which 25 minutes will be related to study specific procedures.

Subjects Patients referred by General practitioners or Otolaryngologists for hearing aid fittings to the offices of two Audiologists who meet the inclusion criteria will be provided with details of the study including a participant information and consent form at their initial evaluation.

Study Procedures Recruitment Patients who satisfy the inclusion criteria will be invited to participate in the study and complete a study consent form.

Allocation Consenting patients will be assigned a study ID and randomized into the Control or Test group using a table of random numbers.

Intervention Process Consenting patients will be randomised using a random number table to have a post-fitting visit between days 21 to 60 after the initial hearing aid fitting with an Audiologist (Control group) or the referring Physician (Test Group). At this visit the audiologist or physician will document the degree of hearing change in specific listening environment/situations as a result of hearing aid use by following the COSI questionnaire. This visit will be for a maximum of 30 minutes.

A follow-up visit of this nature is part of routine clinical practice for the participating audiologist. The physician visit is the novel study intervention after which the patient returns for all subsequent follow-ups with the hearing aid fitting audiologist in keeping with routine clinical practice.

Patient data to be collected

Demographics:

• age, sex

Clinical data:

• degree of hearing loss

Data Analysis The primary indicator of patient satisfaction will be the scored 15-item SADL questionnaire. The Statistical Program for the Social Sciences will be used to undertake a t-test or ANOVA comparison of the mean total SADL questionnaire scores in the Control and Test groups. The secondary outcome measure hearing aid returns, will be assessed by Chi-squared tests of the proportion of returned hearing aids returned in both groups.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Sensorineural hearing loss greater than 25 dB averaged over frequencies 0.5, 1, 2 and 4 KHz; or 2, 3 and 4 KHz on pure tone audiometry in either ear.
* Have used a hearing for up to 21 days after being fitted

Exclusion Criteria:

* Age under 55 years
* Unable to follow doctor/audiologist's instructions
* Previous hearing aid use

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-07; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Amplification in Daily Life questionnaire score | SADL questionnaire completed at patient's final visit or when hearing aid is returned (77-90 days from initial hearing aid fitting)
  Participant determined satisfaction level with the hearing aid based on the Satisfaction with Amplification in Daily Life (SADL) questionnaire score.

SECONDARY OUTCOMES:
Proportion of Hearing aid returned | 77-90 day post fitting
  Participant dissatisfaction with the hearing aid based on the proportion of hearing aids returned

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Nunez, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
We intend to IPD post publication of the study's findings. We estimate that this will be from July 2019
Supporting Information: CSR
Time Frame: From July 2019- June 2020
Access Criteria: By contacting corresponding author in peer reviewed publication.

REFERENCES:
- [Derived] Zhao K, Hambley M, Venema T, Marynewich S, McNeely B, Nunez DA. Effect of Physician Consultation on Satisfaction With Hearing Aid Use: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Jul 1;148(7):630-635. doi: 10.1001/jamaoto.2022.0927. PMID 35588353